CLINICAL TRIAL: NCT03255369
Title: Vertical Exposure to Zika Virus and Its Consequences for Child Neurodevelopment: Cohort Study in Fiocruz/IFF
Brief Title: Vertical Exposure to Zika Virus and Its Consequences for Child Neurodevelopment (ZIKVIRUSIFF)
Acronym: ZIKVIRUSIFF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 52675616.0.0000.5269
Record Dates: First submitted 2017-08-16; First posted 2017-08-21 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2017-08

CONDITIONS: ZIKA VIRUS INFECTION; Child Development; Microcephaly
Keywords: Zika virus; Microcephaly; Child; pregnancy
MeSH Terms: conditions — Zika Virus Infection; Microcephaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Urine and blood for RT-PCR Blood for IgG and IgM Saliva for RT-PCR placenta oral swab for genetic studies fetal tissues stillborn for necropsy CSF and amniotic fluid if affected babies breastmilk
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Child exposed Zika virus proved: child born to mothers with proved zika virus in pregnancy by RT-PCR
  Interventions: Other: Child exposed Zika virus proved
- Child exposed to zika virus suspected: Child born with symptoms similar to babies proved exposed to zika virus but mothers without symptoms or positive RT-PCR
  Interventions: Other: Child exposed Zika virus proved
- Normal Child: Normal child from mothers without Zika (IgG and IgM negative)
  Interventions: Other: Child exposed Zika virus proved

INTERVENTIONS:
Other: Child exposed Zika virus proved — There will be applied Bayley Teste 3rd edition
  Other Names: Child exposed Zika virus suspected

SUMMARY:
The recent increase in the number of cases of congenital microcephaly observed in Brazil is a reason of great concern. This increase occurred a few months after Zika virus (ZIKV) was introduced in the country, which was associated with reports of pregnant women presenting fever and rash illness during pregnancy. Thus, the hypothesis of a relationship between ZIKV infection and microcephaly became plausible. However, studies on the pathophysiology of maternal ZIKV infection, its consequences for the fetus, and the development of severe encephalopathy are still needed. Knowledge about the natural history of vertical transmission and its association with changes in fetal development in early life is still scarce. Studies on factors which determine the severity and clinical evolution, such as inflammatory response mechanisms, viral evolution, and development of serological tests to identify ZIKV infection, are still needed. The Aedes aegypti is responsible for the transmission of various types of viruses of interest to human health. Currently, it is primarily responsible for the transmission of the dengue, chikungunya, and ZIKV in epidemic proportions. In addition, it is not yet known whether there is an interaction between these viruses and whether the interaction can determine the severity of the disease. The aim of this study is to evaluate the natural history of ZIKV disease in two cohorts( pregnant women and children) starting with pregnant women or newborns or evennursing mothers, identifying risk biomarkers, mapping the anti-viral inflammatory response, evaluating the molecular evolution of the virus,which areimportant to determine the mechanisms of vertical viral infection and verify children neurodevelopment from birth to the end of 3rd year of life.

DETAILED DESCRIPTION:
The mais goal of the study is to assess the natural history of vertical ZIKV transmission from pregnancy to the end of third year of life and the existence of risk factors associated with the incidence of clinical and neurological disorders, specially microcephaly.

A longitudinal study will be conducted from gestation to the end of the third year of life, during which ZIKV infection will be the main exposure.

Sample size will be 500 children exposed to zika virus. The sample size was calculated for rare events with basis on the usual microcephaly prevalence in Brazil (2:10.000) and expected increase in the number of cases among pregnant women exposed to ZIKAV.

The study will be conducted at the Fernandes Figueira National Institute for Health of Women and Children (IFF). The pregnant women will be selected in the prenatal care clinic at IFF and in the Family Health Strategy units, at Centro de Saúde Escola Germano Sinval Faria (CDEGSF), which are both from FioCruz/RJ. We also will recruit pregnant woman from clinical family of SMS Rio de Janeiro.

Inclusion criteria The study population will be composed of pregnant women who present symptoms compatible with ZIKAV infection, with skin rash, arthralgia-associated fever, myalgia, non-purulent conjunctivitis, or headache and asymptomatic pregnant women identified at the same time of possibility of exposure. We will include patients with RT- PCR positive.

All pregnant women who are in the prenatal follow up at IFF and CSGSF, irrespective of the gestational age, are elegible as a not exposed in the beginning.

Exclusion criteria Pregnant women with chromosomal abnormalities detected during fetal life or birth will be excluded.

Definition of exposure Given the knowledge that about 80% of ZIKAV infections are asymptomatic, the exposure will be confirmed by the positivity in diagnostic tests (PCR or serological tests). Considering the future availability of serological tests, some strategies will be used to define exposure groups because up to now only the PCR test is available, which remains positive only in the acute phase of the disease.

As described above, the symptomatic women will be referred for infection diagnostic confirmation by RT-PCR , and serologic tests for dengue, chikcungunha, CMV, toxoplasmosis, and rubella.

Women with and without symptoms will have their blood sampled for serological tests in the three trimesters of pregnancy and at birth. Blood samples will be stored in a biorepository for ZIKA serological testing when specific serological tests are available. These sequential samples will also be used to validate serological tests that are in the development stage.

The exposure groups to be compared will be composed with basis on the results of the serological tests. The asymptomatic individuals whose blood samples indicate the presence of Zika infection in the future, will migrate to the group of exposed ones.

The pregnant women in the cohort presenting positive results for specific tests (PCR in the acute phase and serological tests later) will be considered exposed to infection whereas pregnant women with negative results will be considered not exposed.

This second group can be categorized as asymptomatic and symptomatic. The third group will be the normal children born from mothers without zika proved by negative IgG and IgM Each child will be followed for three years from birth onwards.

Outcomes to be analyzed The main outcome will be microcephaly and/or delay in development using Bayley Score 3rd edition at 12, 18 and 24-36 months of age.

The secondary study outcomes will be as follows: pregnancy ultrasounds status, placenta injuries, ocular, hearing, cardiac, nutritional status of children and neurodevelopmental changes from birth to three years old, death in pregnant women, abortion, fetal death, and death during the first three years of life.

Data collection:

The inclusion of pregnant women will occur in the first 24 months of the study. To identify the outcomes, each child will be followed from birth to completion of three years of chronological age. The total study period for data collection will be of 5 years. The study will be conducted in the period Jan 2016 - Mar 2022.

Data will be collected by health professionals who are linked to health services and provide assistance to the study population.

Data on gestation, birth, and the first three years of life will be obtained from an interview with each woman using a questionnaire after appointment. In addition, data for records will be collected in forms prepared for this purpose.

The data collection form (CRF/DCF) will be constructed and validated in all its dimensions among the services. POPs for the study flow diagram and for each procedure and care level will be prepared.

* Socioeconomic characteristics (education, per capita family income, housing conditions, sanitation, and garbage collection); health conditions (co-morbidities).
* History of exposure to ZIKAV: identification of relatives, neighbors, and work colleagues with Zika

Follow up of the study population

Follow up of the pregnant women:

The pregnant women included in the study will be followed in the prenatal clinic, at the Fernandes Figueira National Brazilian Institute for Health of Women and Children.

After inclusion of the pregnant women in the study, consultations will occur monthly, and exams will be performed according the following protocol:

* Fetal ultrasound at each trimester
* Serological exams for Zika, dengue, chikungunya, CMV, toxoplasmosis and rubella each trimester
* PCR for Zika virus if symptomatic pregnant woman
* Prenatal examinations as recommended by the Stork Network from Brazilian Minister of Health
* Prenatal examinations as recommended by the Brazilian Stork Network The amniotic fluid can be collected if indicated by the presence of associated congenital anomalies.

Doppler:

The umbilical cord will be insonated to obtain a sonogram of the umbilical artery and thus assess the pulsatility index (PI), resistance index (RI), and peak systolic velocity (PSV).

Virus detection in serum and other human secretions For detection of virus in patients, RNA is extracted from serum and/or urine (200 ml) using the RTP Pathogen (Stratec Biomedical AG, Birkenfeld, Germany) kit according to the manufacturer's instructions. RNA isolated serves as a template in in real-time /RT-PCRreactions asdescribed by: Lanciotti et al., 2008 e Faye et al., 2013.

Virus detection in serum and other human secretions For genomic sequencing, specific regions of the virus genome will be amplified by the RT-PCR method. The products thusobtained will be purified by agarose gel electrophoresis and then extracted from the gel using the QIAquick Gel Extraction (Qiagen) kit. After extraction, the material will be quantified in agarose gel by comparison between band intensities using the Low DNA Mass Ladder (Life Technologies) standard. The amount needed for sequencing will be forwarded to the Fiocruz sequencing platform. The sequences will be manually edited using the Bioedit (v. 7.0.5.3) program, and the phylogenetic analyses will be performed using the MEGA (v. 5:05) program.

Analysis of the placenta and immunohistochemistry The fresh placentas will be forwarded to the Department of Pathological Anatomy and Cytopathology (DAPC/DPAC) where they will be kept in the refrigerator for up to 48 h. They are described, weighed, and photographed according to the routine for analysis of placenta. Fragments from the chorionic plate, cord, and membranes will be removed and frozen in liquid nitrogen. The placental plate (five areas), cord (at least two areas), and chorion (one fragment) will be fixed in buffered formalin maximum time: 30 h). They will be then cleaved for histological processing and embedded in paraffin.

Phenotypic characterization of placental cells and maternal and umbilical cord blood and child oral swab by flow cytometry Placental fragments will be collected and maintained in sterile DMEM (Sigma; St. Louis, MO, [USA]) culture medium (4 °C) and cleaved into several fragments (thickness: 1-2 mm). After cleavage, they are washed in DMEM and subjected to dissociation cycles in collagenase 1A (Sigma; _) (300 U/mg; in 1% DMEM) enzyme. Dissociation will occur in 6-8 cycles (mild agitation; 37 °C, 10 min each). The cell suspension thusobtained will be centrifuged (1000 rpm; 4 °C; 10 min) and the pellet will be placed /suspended in DMEM with fetal calf serum (FCS; 10%; Sigma; _; 4 °C) to /inactivate /inhibit the collagenase enzyme /action /activity?. The dissociated material will [then] be filtered /in /through?a membrane ([pore diameter:] 70 mm). Then, the cells will be counted in a Neubauer chamber for use in the following procedures. The maternal and umbilical cord blood will be collected in /a blood /an appropriate tube containing EDTA as anticoagulant. The serum will be used for viral detection, and the leukocyte cells will be marked after lysis of red blood cells.\

Necropsy of Fetuses and Stillbirths Histopathological and immunohistochemical exams and imaging morphogenesis study will be performed in brain and other organs from fetuses and stillbirths /in consequence of ZIKAV infection. Besides the usual histological processing in paraffin, the other organs will be frozen and submitted to extraction of genetic material and investigation of viral RNA. The eyeball will also be analyzed to evaluate possible ocular changes.

Follow-up of newborns:

Newborns will be followed until 3 years of age in the outpatient clinic at IFF, whose routine includes at least 6 visits in the first year, 4 visits/year in the second and third years. A multidisciplinary outpatient clinic will be established in both Unit of Infectious Diseases in Pediatrics and Pediatric Outpatient Clinic to follow the cohort of children with chance of vertical exposure to the ZIKA virus. The outpatient clinic will have medical personnel, and professionals in the areas of physical therapy, phonoaudiology, psychology, and social service. The medical team will be responsible for following the patients, in collaboration with specialties as neurology, pediatric cardiology and ophthalmology, and medical genetics service. Whenever necessary, admission of these patients to establish [either] the diagnosis or initial approach -{of the case} will occur in the DIPe ward.

The initial evaluation as recommended for patients either known to be exposed to the virus or with microcephaly will consist of the following exams and/or evaluations: neurological, ocular, hearing, EEG if necessary, ECG, cord blood for RT-PCR and IgM. Anthropometric data and physical examination of the newborn infant, with emphasis on precise measurement of head circumference using the Intergrowth Curve (2014) as a reference, according to gestational age and patient gender. Evaluation by the Genetics to detect dysmorphic characteristics or congenital anomalies that can compromise /affect other organs.

Imaging exams:

1. transfontanelle sonography (USTF), as first choice
2. cranial tomography (CT) without contrast, if TF is not technically possible
3. Abdominal ultrasound
4. Echocardiogram
5. Brain magnetic resonance imaging, when indicated. g) Newborn Hearing Screening (TAN):

1. Evoked optoacoustic emissions (EOAE); 24-48 h of life 2. Auditory Evoked Potential of Brain Stem (PEATE/ABR): up to 1 month of life in children with microcephaly. In case of failure, retesting must be done within 30 days. In case of retest failure, forward [the NB] immediately [to _].

h) Ocular Neonatal Screening (TON):

1. Inspection and Testing of retinal Red Reflection.
2. Eye Fund exam (fundoscopy)
3. Documentation with RetCam

In the subsequent consultations, the clinical follow up, PC measurement, development evaluation (including early stimulation) by physical therapy, and morbidity and mortality evaluation will be maintained. In the first year of life, PEATE will be performed every three months. The subsequent clinic visits will occur monthly until 6 months of age, every two months in the period 6-12 months, and every three months until three years [of life]. The ophthalmologic evaluation (funduscopic examination) will be held every return.

The neurological follow up will depend on the initial condition of the patient. Patients without microcephaly will be evaluated at birth, 30 days, and 2, 4, 6, 9, 12, 18, 24, and 36 months. Patients with microcephaly will be evaluated at birth, 30 days, and every 2 or 3 months, or more frequently if necessary.

Evaluation of motor development will be done by the Dubowitz examination (in the first 72 h), Alberta Infant Motor Scale (AIMS; every three months until the child walk or complete 18 months of life), and Bayley Test-3rd edition at 12,18 and between 12-36 months of age.

Evaluation of language development will be performed at 12, 24, and 36 months, with regard to possible effects on the neurodevelopment, cognitive development, and language skills.

ELIGIBILITY:
Inclusion Criteria:

The study population will be composed of pregnant women who present symptoms compatible with ZIKAV infection, with skin rash, arthralgia-associated fever, myalgia, non-purulent conjunctivitis, or headache and asymptomatic pregnant women identified at the same time of possibility of exposure. We will include patients with RT- PCR positive.

All pregnant women who are in the prenatal follow up at IFF and CSGSF, irrespective of the gestational age, are elegible as a not exposed in the beginning.

Children born during the outbreak by mothers with confirmed infection, suspected infection and normal pregnancy

Exclusion Criteria:

Pregnant women with chromosomal abnormalities detected during fetal life or birth will be excluded.

-

Ages: 2 Days to 3 Years | Sex: All
Age Groups: Child
Study Population: The exposure will be confirmed by the positivity in diagnostic tests (PCR or serological tests).
  Women with and without symptoms will have theirblood sampled for serological tests in the three trimesters of pregnancy and at birth.
  The pregnant women in the cohort presenting positive results for specifictests (PCR in the acute phase and serological tests later) will be considered exposed to infection whereas pregnant women with negative results will be considered not exposed.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01-02 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Microcephaly and/or delay in development | 36 months of age
  Microcephaly at birth or delay in development in Bayley test 3rd edition at 12, 18 and between 24-36 months of age

SECONDARY OUTCOMES:
ocular injury and cognitive disorder in Bayley Test 3rd edition | 36 months of age
  ocular injury in eye exam by indirect ophtalmoscopia registe by RetCam associated with cognitive disorder
Hearing injury and language delay in Bayley Test 3rd edition | 36 monthsof age
  deaphness or BERA abnomalities associated to language disorder

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Moreira, MD, Principal Investigator — Fundação Oswaldo Cruz
Locations (1):
- Instituto Fernandes Figueira/Fiocruz, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
we will share the data with Brazilian Minister of Health, WHO and European ZikaPlane consortium
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: 3 years
Access Criteria: only the principal investigator

REFERENCES:
- [Background] Brasil P, Pereira JP Jr, Moreira ME, Ribeiro Nogueira RM, Damasceno L, Wakimoto M, Rabello RS, Valderramos SG, Halai UA, Salles TS, Zin AA, Horovitz D, Daltro P, Boechat M, Raja Gabaglia C, Carvalho de Sequeira P, Pilotto JH, Medialdea-Carrera R, Cotrim da Cunha D, Abreu de Carvalho LM, Pone M, Machado Siqueira A, Calvet GA, Rodrigues Baiao AE, Neves ES, Nassar de Carvalho PR, Hasue RH, Marschik PB, Einspieler C, Janzen C, Cherry JD, Bispo de Filippis AM, Nielsen-Saines K. Zika Virus Infection in Pregnant Women in Rio de Janeiro. N Engl J Med. 2016 Dec 15;375(24):2321-2334. doi: 10.1056/NEJMoa1602412. Epub 2016 Mar 4. PMID 26943629
- [Background] Chimelli L, Melo ASO, Avvad-Portari E, Wiley CA, Camacho AHS, Lopes VS, Machado HN, Andrade CV, Dock DCA, Moreira ME, Tovar-Moll F, Oliveira-Szejnfeld PS, Carvalho ACG, Ugarte ON, Batista AGM, Amorim MMR, Melo FO, Ferreira TA, Marinho JRL, Azevedo GS, Leal JIBF, da Costa RFM, Rehen S, Arruda MB, Brindeiro RM, Delvechio R, Aguiar RS, Tanuri A. The spectrum of neuropathological changes associated with congenital Zika virus infection. Acta Neuropathol. 2017 Jun;133(6):983-999. doi: 10.1007/s00401-017-1699-5. Epub 2017 Mar 22. PMID 28332092
- [Background] Halai UA, Nielsen-Saines K, Moreira ML, de Sequeira PC, Junior JPP, de Araujo Zin A, Cherry J, Gabaglia CR, Gaw SL, Adachi K, Tsui I, Pilotto JH, Nogueira RR, de Filippis AMB, Brasil P. Maternal Zika Virus Disease Severity, Virus Load, Prior Dengue Antibodies, and Their Relationship to Birth Outcomes. Clin Infect Dis. 2017 Sep 15;65(6):877-883. doi: 10.1093/cid/cix472. PMID 28535184
- [Result] Zin AA, Tsui I, Rossetto J, Vasconcelos Z, Adachi K, Valderramos S, Halai UA, Pone MVDS, Pone SM, Silveira Filho JCB, Aibe MS, da Costa ACC, Zin OA, Belfort R Jr, Brasil P, Nielsen-Saines K, Moreira MEL. Screening Criteria for Ophthalmic Manifestations of Congenital Zika Virus Infection. JAMA Pediatr. 2017 Sep 1;171(9):847-854. doi: 10.1001/jamapediatrics.2017.1474. PMID 28715527
- [Derived] Tiene SF, Cranston JS, Nielsen-Saines K, Kerin T, Fuller T, Vasconcelos Z, Marschik PB, Zhang D, Pone M, Pone S, Zin A, Brickley E, Orofino D, Brasil P, Adachi K, da Costa ACC, Lopes Moreira ME. Early Predictors of Poor Neurologic Outcomes in a Prospective Cohort of Infants With Antenatal Exposure to Zika Virus. Pediatr Infect Dis J. 2022 Mar 1;41(3):255-262. doi: 10.1097/INF.0000000000003379. PMID 35144270